CLINICAL TRIAL: NCT00005669
Title: Effects of Metformin on Energy Intake, Energy Expenditure, and Body Weight in Overweight Children With Insulin Resistance
Brief Title: Metformin to Treat Obesity in Children With Insulin Resistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jack Yanovski, M.D. (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Jack Yanovski, M.D., Chief, Section on Growth and Obestiy, PDEGEN, NICHD, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000134; 00-CH-0134 (Other: NIH Clinical Center)
Record Dates: First submitted 2000-05-19; First posted 2000-05-22 (Estimated); Results first posted 2011-04-07 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-04

CONDITIONS: Hyperinsulinemia; Obesity
Keywords: Child; Body Fat; Food Intake; Diabetes Mellitus; Dyslipidemia; Vitamin B12; Childhood Obesity
MeSH Terms: conditions — Hyperinsulinism; Obesity; Diabetes Mellitus; Dyslipidemias; Pediatric Obesity | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Metformin HCL (Active Comparator): Subjects receive metformin plus a weight loss program
  Interventions: Drug: Metformin HCL
- 2 - Placebo (Placebo Comparator): Subjects receive placebo plus a weight loss program
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin HCL — Medication studied for ability to alter body weight and body composition.
  Arms: 1 - Metformin HCL
Drug: Placebo — Control capsules for metformin
  Arms: 2 - Placebo

SUMMARY:
This study will examine the safety and effectiveness of the medicine metformin to help overweight children control their food intake, weight, insulin, cholesterol, and triglyceride (blood fat) levels. Obesity and high insulin levels can lead to high blood pressure, diabetes, high cholesterol and triglyceride levels and heart disease. Metformin-approved by the Food and Drug Administration to treat adults with type 2 diabetes mellitus-helps lower insulin levels and may control weight gain in adults.

Overweight children 6 to 11 years old who are in general good health may be eligible for this study. Children will be studied at the National Institutes of Health in Bethesda, Maryland. Candidates will have a medical history and physical examination and fasting blood test, and will provide a 7-day record of their food intake as part of the screening process. Those enrolled will be randomly assigned to receive either metformin or placebo (a look-alike tablet with no active medicine) twice a day for a six month period. After the 6 month study period, all children will be offered the opportunity to take metformin for another 6 months.

Participants will be hospitalized for 2-3 days for the following procedures: history and physical examination; fasting blood test; several urine collections; X-ray studies to determine bone age and amount of body fat and muscle; magnetic resonance imaging (MRI) scan to measure body fat; "hyperglycemic clamp study" to evaluate insulin resistance; food intake testing; nutrition consultation; resting metabolic rate; and a "doubly labeled water" test.

For the hyperglycemic clamp study, a catheter (thin flexible tube) is inserted into a vein in each arm. A sugar solution is given through one tube and blood samples are drawn every 5 minutes through the other to measure insulin. For the food intake testing, the child is asked about his or her hunger level, then given various foods he or she may choose to eat, then questioned again at various intervals both during and after finishing eating about his or her hunger level. The doubly labeled water study involves drinking "heavy water" (water which is enriched to have special kinds of hydrogen and oxygen). Urine specimens are collected 2, 3 and 4 hours after drinking the water. The child also drinks a special milk shake called a Scandishake and repeats the calorie intake and hunger study. (Two food intake studies are done on separate days.) One week after the heavy water test, additional urine samples are collected one week later.

After completing the tests, the child will begin treatment with metformin or placebo, plus a daily vitamin tablet. Participants will be followed once a month with a brief history and physical examination, including a blood test. After 6 months, all of the tests described above will be repeated. All children who complete the second round of tests-both those who took metformin and those who took placebo-will be offered metformin for an additional 6 months and will be seen once a month for follow-up evaluations. Parents will not be told which children received metformin and which received placebo until all children in the study complete the first 6 months of the trial.

DETAILED DESCRIPTION:
The prevalence of overweight and obesity in children and adolescents in the United States has doubled during the past 20 years. Obesity is closely linked with development of insulin resistance and other mediators of unfavorable cardiovascular risk, such as hypertension and dyslipidemia. These obesity-related risk factors often first appear during childhood. Since obese children tend to become obese adults, such children are at increased risk for persistence of these abnormalities into adulthood and for the early occurrence of obesity-related morbidity and mortality. Obesity-related insulin resistance is also largely responsible for the recently documented rise in the incidence of Type 2 diabetes in youth. To date, there is no FDA-approved pharmacotherapy for children with obesity and insulin resistance. Metformin is a medication approved for use in adults with Type 2 diabetes that is unique in that it promotes weight loss and improves features of the insulin resistance syndrome. Preliminary studies suggest that metformin may promote weight loss in obese non-diabetic children. However, the mechanism of metformin-induced weight loss has not been elucidated. We propose to evaluate the safety, tolerability, efficacy and mechanism of metformin-induced weight loss in obese, hyperinsulinemic children aged 6-12.99 years. We will conduct a six-month randomized, double blind placebo-controlled trial of metformin. All study participants will receive nutritional consultation and advice on appropriate diet. We will study the effects of metformin on weight, food intake, energy expenditure, insulin sensitivity, and lipids. At the end of the six-month placebo-controlled trial, all subjects will be offered metformin in an open label phase for an additional six months.

ELIGIBILITY:
* INCLUSION CRITERIA:

Good general health.

Age greater than or equal to 6 and less than 13 years.

Pre-pubertal or having at most early puberty (breast Tanner I, II or III for girls, testes size less than or equal to 8 mL for boys).

Hyperinsulinemia, defined as fasting insulin concentration greater than or equal to 15 mIU/mL. The insulin level must be greater than or equal to 15 at either the NIH Clinical Center lab or the NIDDK lab at PIMC in Phoenix.

Obesity, defined as body mass index greater than or equal to 95th percentile determined by NHANES I age and sex specific data.

Subjects must have fasting plasma glucose less than 126 mg/dl

Subjects must have glycosylated hemoglobin (HgbA1C) of less than or equal to 6.5%.

Females who begin menstruating (or who are at risk for pregnancy) during the study must have a negative pregnancy test and must use an effective method of contraception if they are engaging in sexual intercourse.

EXCLUSION CRITERIA:

Baseline creatinine greater or equal to 1.0 mg/dl.

Significant cardiac or pulmonary disease likely to or resulting in hypoxia or decreased perfusion.

Hepatic disease with elevated liver function tests (ALT or AST) greater than or equal to 1.5 the upper limits of normal.

An alcohol history concerning for development of hepatic toxicity.

Pregnancy.

Evidence for Type 2 diabetes, including fasting plasma glucose greater than or equal to 126 mg/dl or HgbA1C greater than 6.5%.

Weight loss of greater than 2% of bodyweight within the past 6 months.

Presence of other endocrinologic disorders leading to obesity (e.g. Cushing's Syndrome).

Individuals who have, or whose parent or guardians have current substance abuse or a psychiatric disorder or other condition that, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study.

Recent use (within six months) of anorexiant medications.

Individuals receiving medical treatment other than diet for hypertension or dyslipidemia.

Individuals with evidence of precocious puberty.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2000-05; Primary Completion 2009-08 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, MD, PhD, Principal Investigator — NICHD, NIH
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bao W, Srinivasan SR, Wattigney WA, Berenson GS. Persistence of multiple cardiovascular risk clustering related to syndrome X from childhood to young adulthood. The Bogalusa Heart Study. Arch Intern Med. 1994 Aug 22;154(16):1842-7. PMID 8053753
- [Background] Wilson DM, Abrams SH, Aye T, Lee PD, Lenders C, Lustig RH, Osganian SV, Feldman HA; Glaser Pediatric Research Network Obesity Study Group. Metformin extended release treatment of adolescent obesity: a 48-week randomized, double-blind, placebo-controlled trial with 48-week follow-up. Arch Pediatr Adolesc Med. 2010 Feb;164(2):116-23. doi: 10.1001/archpediatrics.2009.264. PMID 20124139
- [Background] Melnik TA, Rhoades SJ, Wales KR, Cowell C, Wolfe WS. Overweight school children in New York City: prevalence estimates and characteristics. Int J Obes Relat Metab Disord. 1998 Jan;22(1):7-13. doi: 10.1038/sj.ijo.0800537. PMID 9481594
- [Derived] Manoli I, Sysol JR, Head PE, Epping MW, Gavrilova O, Crocker MK, Sloan JL, Koutsoukos SA, Wang C, Ktena YP, Mendelson S, Pass AR, Zerfas PM, Hoffmann V, Vernon HJ, Fletcher LA, Reynolds JC, Tsokos MG, Stratakis CA, Voss SD, Chen KY, Brown RJ, Hamosh A, Berry GT, Chen XS, Yanovski JA, Venditti CP. Lipodystrophy in methylmalonic acidemia associated with elevated FGF21 and abnormal methylmalonylation. JCI Insight. 2024 Feb 22;9(4):e174097. doi: 10.1172/jci.insight.174097. PMID 38271099
- [Derived] Han JC, Reyes-Capo DP, Liu CY, Reynolds JC, Turkbey E, Turkbey IB, Bryant J, Marshall JD, Naggert JK, Gahl WA, Yanovski JA, Gunay-Aygun M. Comprehensive Endocrine-Metabolic Evaluation of Patients With Alstrom Syndrome Compared With BMI-Matched Controls. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2707-2719. doi: 10.1210/jc.2018-00496. PMID 29718281
- [Derived] Adeyemo MA, McDuffie JR, Kozlosky M, Krakoff J, Calis KA, Brady SM, Yanovski JA. Effects of metformin on energy intake and satiety in obese children. Diabetes Obes Metab. 2015 Apr;17(4):363-70. doi: 10.1111/dom.12426. Epub 2015 Jan 11. PMID 25483291
- [Derived] Yanovski JA, Krakoff J, Salaita CG, McDuffie JR, Kozlosky M, Sebring NG, Reynolds JC, Brady SM, Calis KA. Effects of metformin on body weight and body composition in obese insulin-resistant children: a randomized clinical trial. Diabetes. 2011 Feb;60(2):477-85. doi: 10.2337/db10-1185. Epub 2011 Jan 12. PMID 21228310
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2000-CH-0134.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited subjects from 2000 through 2008. Obese children (BMI 95th percentile or greater), aged 6-12y, were recruited through newspaper advertisements and letters to physicians, and were eligible if they had fasting hyperinsulinemia, (insulin at least 15mU/mL. Following an outpatient screen, participants were admitted for assessments.
Pre-assignment Details: Children were excluded if they had impaired fasting glucose or were diabetic, had significant renal, hepatic, cardiac or pulmonary disease, or presence of other endocrinologic disorders leading to obesity, had used prescription or non-prescription weight loss agents, or reported >2% body weight loss in the preceding 6 months.
Groups:
- Metformin Plus Weight Reduction Counseling: Subjects receive increasing doses of metformin to the maximum of 2000 mg per day (metformin supplied as 250 mg capsules administered with breakfast and dinner) plus a weight loss program
- Placebo Plus Weight Reduction Counseling: Subjects receive increasing doses of placebo to the maximum of 2000 mg per day (placebo supplied as 250 mg capsules administered with breakfast and dinner) plus a weight loss program
Period: Overall Study
Arm/Group | Metformin Plus Weight Reduction Counseling | Placebo Plus Weight Reduction Counseling
Started | 53 | 47
Completed | 45 | 40
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin Plus Weight Reduction Counseling | Placebo Plus Weight Reduction Counseling | Total
Number analyzed (Participants) | 53 | 47 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 53 | 47 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (1.6) | 10.4 (1.4) | 10.2 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 23 | 17 | 40
Region of Enrollment [Number; unit: participants]
  United States | 53 | 47 | 100

OUTCOME MEASURES:

1. Primary Outcome: Changes in Body Weight as Determined by Body Mass Index-standard Deviation Score (BMI-SDS).
Description: Change in Body Mass Index standard deviation score (BMI-SDS) determined using tables created by the CDC in 2000. BMI-SDS is a unitless transformation of the body mass index (measured in kg divided by the squared height in meters) using the L M S method. Possible values range from -3 to +3. See http://www.cdc.gov/growthcharts/percentile_data_files.htm for details.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Metformin Plus Weight Reduction Counseling | Placebo Plus Weight Reduction Counseling
Number analyzed (Participants) | 53 | 47
Units on a scale | -0.11 [-0.16 to -0.05] | -0.07 [-0.12 to -0.01]

2. Secondary Outcome: Change in Body Weight as Determined by BMI
Description: Change in body weight as determined by body mass index (kg/m2)
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: kg/m2
Arm/Group | Metformin Plus Weight Reduction Counseling | Placebo Plus Weight Reduction Counseling
Number analyzed (Participants) | 53 | 47
kg/m2 | -0.78 [-1.54 to -0.01] | 0.32 [-0.54 to 1.18]

3. Secondary Outcome: Change in Body Weight
Description: Change in body weight (kg)
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Metformin Plus Weight Reduction Counseling | Placebo Plus Weight Reduction Counseling
Number analyzed (Participants) | 53 | 47
kg | 1.47 [-0.31 to 3.24] | 4.85 [2.84 to 6.85]

4. Secondary Outcome: Change in Body Fat by DEXA
Description: Change in body fat mass by Dual Energy X-Ray Absorptiometry (kg)
Time Frame: 6 months
Population: ITT, multiple imputation model for missing data under a missing-at-random assumption
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Metformin Plus Weight Reduction Counseling | Placebo Plus Weight Reduction Counseling
Number analyzed (Participants) | 53 | 47
kg | 0.48 [-0.80 to 1.76] | 1.88 [0.44 to 3.31]

5. Secondary Outcome: Change in Body Fat by Bod Pod
Description: Change in body fat mass measured by air displacement plethysmography (kg)
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Metformin Plus Weight Reduction Counseling | Placebo Plus Weight Reduction Counseling
Number analyzed (Participants) | 53 | 47
kg | -1.51 [-4.56 to 1.54] | 1.81 [-1.64 to 5.25]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Pharmacist-administered comprehensive structured questionnaire at baseline and follow-up timepoints plus case report forms with specific questions related to expected toxicities of metformin.
Arm/Group | Metformin Plus Weight Reduction Counseling | Placebo Plus Weight Reduction Counseling
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/47
Other Adverse Events (participants affected / at risk) | 48/53 | 46/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin Plus Weight Reduction Counseling (N=53) | Placebo Plus Weight Reduction Counseling (N=47)
Nausea (Gastrointestinal disorders) | 28 (55) | 17 (18)
Liquid Stools (Gastrointestinal disorders) | 22 (34) | 8 (8)
Vomiting (Gastrointestinal disorders) | 22 (36) | 10 (10)
Bloating (Gastrointestinal disorders) | 13 (20) | 6 (7)
Increased Bowel Movements (Gastrointestinal disorders) | 22 (25) | 11 (13)
Fatigue (General disorders) | 20 (29) | 7 (10)
Decreased Happiness (General disorders) | 14 (14) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No